CLINICAL TRIAL: NCT03600792
Title: Whole Exome Sequencing in Prenatal Diagnosis of Agenesis of the Corpus Callosum
Acronym: EXACC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI18011J
Record Dates: First submitted 2018-06-10; First posted 2018-07-26 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Fetal Agenesis of the Corpus Callosum (ACC)
Keywords: Agenesis of the corpus callosum; whole exome sequencing; prenatal diagnosis
MeSH Terms: conditions — Agenesis of Corpus Callosum | interventions — Exome Sequencing

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: whole exome sequencing (WES) — WES analysis will be performed in the "UF de Génomique du Développement" (APHP, Pitié-Salpêtrière hospital), using DNA extracted from amniotic fluid for the foetus (also used for chromosomal studies) and DNA extracted from peripheral blood for both parents. There will be no supplemental invasive sampling for this study. The result of WES will be returned during a consultation with the geneticist and the associated prognosis will be explained in case of molecular diagnosis

SUMMARY:
Agenesis of the corpus callosum (ACC) is one of the most frequent cerebral malformations and is now diagnosed prenatally in most cases. Prenatal counseling is then challenging because of uncertain neurodevelopmental outcome, depending on the genetic cause of ACC. Our purpose is to evaluate the feasibility of sequencing known genes responsible for ACC by whole exome sequencing (WES) in trio (fetus and both parents) when ACC is diagnosed during the pregnancy, in order to provide complete and loyal information on the intellectual prognosis for the fetus.

DETAILED DESCRIPTION:
Agenesis of the corpus callosum (ACC) is one of the most frequent cerebral malformations. The neurodevelopmental outcome of patients with ACC is extremely variable, ranging from normal intelligence to severe intellectual disability (ID). When ACC is discovered during the prenatal period, prenatal counseling is challenging because of this uncertain neurodevelopmental outcome. Currently, only chromosomal analyses are performed in cases of prenatal diagnoses, which are expected to bring the diagnosis in only few cases. No molecular studies of genes implied in ACC with or without ID are performed. Then, the couples are in the difficult situation of continuing or interrupting the pregnancy without complete information about the aetiology of ACC.

All patients will have a consultation with an obstetrician and consultations with a paediatric neurologist and a geneticist. The geneticist will explain WES and its issues. Both parents will have to provide informed consent for the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* ACC diagnosed prenatally during the 2nd trimester of pregnancy, confirmed by ultrasound by a referee
* Fetal sample (amniotic fluid, 10 ml) et blood samples of both parents (2 tubes of 5 ml EDTA)
* Covered by social security
* Written consent obtain for routine and research genetic analysis

Exclusion Criteria:

* Refusal to participate from one or both parents
* Pregnancies obtained with gamete donation (trio sequencing not feasible)
* If one parent is not available (trio sequencing not feasible)
* Inability to understand the given information
* One or both parents under juridical protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 trios (fetus and both parents) with confirmed diagnosis of fetal ACC during the 2nd or 3rd trimesters of pregnancy and who wish to perform molecular prenatal sequencing by WES.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-10-19 (Actual); Study Completion 2019-10-19 (Actual)

PRIMARY OUTCOMES:
Technical success | 5th week post diagnosis
  Rate of technical success

SECONDARY OUTCOMES:
Genetic diagnosis | 5th week post diagnosis
  Rate of genetic diagnoses
Technical failure | up to 4 months
  Rate of technical failures
Delay to genetic diagnosis Result | up to 4 months
  Delay between the ACC diagnosis and genetic sequencing known genes responsible for ACC
Parents decision to continue pregnancy | up to 4 months
  Number of continued pregnancies
Parents decision to interrupt pregnancy | up to 4 months
  Number of interrupted pregnancies

CONTACTS AND LOCATIONS:
Overall Officials: Héron Delphine, MD, Principal Investigator — APHP
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided